CLINICAL TRIAL: NCT07306676
Title: Symptoms of Post-traumatic Stress Disorder Complicating Spontaneous Abortion
Brief Title: Post-traumatic Stress Disorder in Spontaneous Abortion
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, PhD, MD, Jagiellonian University
Other Study IDs: 118.0043.1.343.2025
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Spontaneous Abortion
Keywords: Spontaneous Abortion; PTSD
MeSH Terms: conditions — Abortion, Spontaneous; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women who experienced a spontaneous miscarriage during the first trimester of pregnancy: Recruitment will take place at the Department of Endocrinology and Gynecology at the University Hospital in Kraków, located at ul. Kopernika 23, 31-501 Kraków, and at the Department of Gynecology and Gynecological Oncology NSSU, located at Jakubowskiego 2, 30-688 Kraków. The study plans to enroll 200 women aged 18 to 45 years who have been hospitalized due to a spontaneous miscarriage.
  Interventions: Diagnostic Test: Impact of Event Scale - Revised (IES-R) questionnaire; Diagnostic Test: Posttraumatic Stress Disorder Checklist - Specific (PCL-S) questionnaire; Diagnostic Test: Trauma Recovery Measure (TRM) questionnaire

INTERVENTIONS:
Diagnostic Test: Impact of Event Scale - Revised (IES-R) questionnaire — The test consists of 22 questions that relate to the respondent's feelings, behaviors, and thoughts concerning the traumatic event over the past seven days. For each question, respondents will indicate one of five responses that best reflects their experience:
  0 - Not at all
  1. - A little
  2. - Moderately
  3. - Often
  4. - Very often
  Upon completion of all questions and totaling the points, the scale for symptoms is classified as follows:
  0-23 points: No or mild symptoms 24-32 points: A significant number of symptoms 33 points or more: Most symptoms characteristic of PTSD.
Diagnostic Test: Posttraumatic Stress Disorder Checklist - Specific (PCL-S) questionnaire — This test includes 17 questions related to the behaviors and feelings of the respondent over the past month. Each question is answered using a 5-point scale with assigned points:
  Not at all - 1 point Sometimes - 2 points Moderately often - 3 points Often - 4 points Very often - 5 points
  After totaling the points, they are classified as follows:
  17-29 points: No or few PTSD symptoms 30-44 points: Moderate to moderately high PTSD symptoms 45-85 points: Numerous PTSD symptoms.
Diagnostic Test: Trauma Recovery Measure (TRM) questionnaire — The stage of recovery is presented based on the distance of the score from the mean. There are three possible stages of recovery:
  * Early Stage of Recovery: Less than 1 standard deviation below the mean (total score of 31 or fewer).
  * Middle Stage of Recovery: Total score ranging from 32 to 61.
  * Late Stage of Recovery: More than 1 standard deviation above the mean (total score of 62 or more).

SUMMARY:
The objective of this questionnaire-based study is to prospectively assess the prevalence of post-traumatic stress disorder (PTSD) symptoms in a population of women who have experienced a spontaneous miscarriage during the first trimester of pregnancy. The investigation into the prevalence of PTSD symptoms will assist in better identifying women who may benefit from early psychological intervention.

DETAILED DESCRIPTION:
A questionnaire-based study will be conducted with prospective inclusion of participants, based on the analysis of medical documentation and self-administered questionnaires. The following questionnaires are proposed for use:

i. Impact of Event Scale - Revised (IES-R) is a 22-item test that measures the level of stress and anxiety resulting from traumatic events. It is utilized as a screening tool in diagnosing post-traumatic stress disorder (PTSD). The test consists of 22 questions that relate to the respondent's feelings, behaviors, and thoughts concerning the traumatic event over the past seven days. For each question, respondents will indicate one of five responses that best reflects their experience: 0 - Not at all

1. - A little
2. - Moderately
3. - Often
4. - Very often

Upon completion of all questions and totaling the points, the scale for symptoms is classified as follows:

0-23 points: No or mild symptoms 24-32 points: A significant number of symptoms 33 points or more: Most symptoms characteristic of PTSD. The questionnaire will be completed during hospitalization.

ii. Posttraumatic Stress Disorder Checklist - Specific (PCL-S) is a 17-item test designed to detect symptoms of PTSD resulting from a specific traumatic event. This test includes 17 questions related to the behaviors and feelings of the respondent over the past month. Each question is answered using a 5-point scale with assigned points: Not at all - 1 point Sometimes - 2 points Moderately often - 3 points Often - 4 points Very often - 5 points

After totaling the points, they are classified as follows:

17-29 points: No or few PTSD symptoms 30-44 points: Moderate to moderately high PTSD symptoms 45-85 points: Numerous PTSD symptoms. The questionnaire will be completed during a routine follow-up visit at the outpatient clinic eight weeks post-discharge from the hospital.

iii. Trauma Recovery Measure (TRM) is a 15-item tool designed to assess trauma and the recovery process. It enables a structured evaluation of the multifaceted impact of trauma on an individual, facilitating the adjustment of support and intervention strategies.

The TRM provides a total score as well as three subscale scores that assess the cognitive aspects of the individual following the experience of traumatic events. The three subscales within the TRM include:

* Validation: This subscale measures the acceptance and self-acceptance of the trauma survivor as they are, despite the traumatic experience, and evaluates the development of internal worth and dignity.
* Liberation: This subscale assesses the survivor's ability to free themselves from control, entrapment, and/or oppression caused by the trauma, and their capacity to live in a way that allows them to feel empowered and confident in making positive decisions for themselves and others.
* Positive Self: This subscale measures the presence of positive cognitive aspects that generate feelings of care, compassion, and/or kindness.

The stage of recovery is presented based on the distance of the score from the mean. There are three possible stages of recovery:

* Early Stage of Recovery: Less than 1 standard deviation below the mean (total score of 31 or fewer).
* Middle Stage of Recovery: Total score ranging from 32 to 61.
* Late Stage of Recovery: More than 1 standard deviation above the mean (total score of 62 or more).

The questionnaire will be completed during a routine follow-up visit at the outpatient clinic eight weeks post-discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous abortion
* gestational age up to 14 weeks.

Exclusion Criteria:

* none

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The prospective survey study will include women receiving treatment in the Department of Endocrinology and Gynecology, as well as the Department of Gynecology and Gynecological Oncology at the University Hospital in Kraków, due to spontaneous abortion diagnosed by the 14th week of gestation. The study plans to enroll 200 women aged 18 to 45 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of Event Scale - Revised (IES-R) score | up to 3 months
  The score obtained from the Impact of Event Scale - Revised (IES-R) questionnaire has a scoring range of 0 to 88 points, with symptom classification according to the following scheme: - 0-23 points: No or mild symptoms - 24-32 points: A significant number of symptoms - 33 points or more: Most symptoms characteristic of PTSD.
Posttraumatic Stress Disorder Checklist - Specific (PCL-S) score | up to 3 months
  The score obtained from Posttraumatic Stress Disorder Checklist - Specific (PCL-S) questionnaire has a scoring range of 17-85 points, with symptom classification according to the following scheme: - 17-29 points: No or few PTSD symptoms - 30-44 points: Moderate to moderately high PTSD symptoms - 45-85 points: Numerous PTSD symptoms.
Trauma Recovery Measure (TRM) score | up to 3 months
  The stage of recovery is presented based on the distance of the score from the mean. There are three possible stages of recovery: - Early Stage of Recovery: Less than 1 standard deviation below the mean (total score of 31 or fewer). - Middle Stage of Recovery: Total score ranging from 32 to 61. - Late Stage of Recovery: More than 1 standard deviation above the mean (total score of 62 or more).

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Gawron, PhD, MD, Study Director — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Krakow, Malopolska, Poland